CLINICAL TRIAL: NCT03541876
Title: Data Collection for the Creation of the French Pediatric Helicobacter Pylori Observatory
Brief Title: French Pediatric Helicobacter Pylori Observatory
Acronym: GFHPP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0058
Record Dates: First submitted 2018-04-23; First posted 2018-05-31 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Helicobacter Pylori Infection
Keywords: children; treatment; observatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — gastric biopsy for histological analysis, culture of bacteria and Polymerase Chain Reaction (PCR)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children with H. pylori infection
  Interventions: Other: Collection of data

INTERVENTIONS:
Other: Collection of data — The following data will be collected by the physician :
  sociodemographic profile (age, sex, country of birth of child and parents); clinical manifestations; endoscopic aspects (esophagus, duodenum, stomach); different methods of diagnosis of infection; different primary and secondary bacterial resistance profiles ; different first and second line therapeutic combinations; different first and second line bacterial eradication rates ; different signs of side effects and tolerance of first and second line treatments; different methods of bacterial eradication control.

SUMMARY:
Helicobacter pylori is a major human pathogen associated with significant morbidity. The treatment oriented by the antibiogram or PCR (Polymerase Chain Reaction) should be privileged in children. However, the optimal treatment for the eradication of pediatric H. pylori infection is still not established.

No French consensus conference on the management of H. pylori infection in children taking into account the epidemiological data available for this infection has been published. The description of diagnostic and therapeutic management procedures has not yet been specifically described according to the country of birth of children. The main objective is to collect data enabling the establishment of a French observatory of Helicobacter pylori in children in order to provide a national database.

ELIGIBILITY:
Inclusion Criteria:

* Child with confirmed H. pylori infection by direct diagnostic methods after periendoscopic gastric biopsies
* Age < 18
* No opposition of at least one of the 2 parents to the use of health data for research purposes

Exclusion Criteria:

* Child with confirmed H. pylori infection by indirect diagnostic methods

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with confirmed diagnosis of H. pylori infection
Sampling Method: Non-Probability Sample
Enrollment: 1201 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of H. pylori infection | at inclusion
  Child with confirmed H. pylori infection by direct diagnostic methods (Histology, Bacterial culture, PCR) on perendoscopic gastric biopsies
Age | at inclusion
Sex | at inclusion
Country of birth | at inclusion
Clinical symptoms | at inclusion, 3 and 6 months
Microbiological diagnosis | at inclusion, 3 and 6 months
Endoscopic diagnosis | at inclusion, 3 and 6 months
Rates of bacterial resistance profiles | at inclusion, at 3 and 6 months
antibiotic therapy | at inclusion, 3 and 6 months
Bacterial eradication rates | 3 and 6 months
Side effects and tolerance of first and second line treatments | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Kalach, PR, Principal Investigator — Lille Catholic University
Locations (1):
- Lille Catholic University, Lille, France